CLINICAL TRIAL: NCT01028729
Title: A Study of Endostar in Combination With Chemotherapy Followed by Endostar Maintenance Therapy in Patients With Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Endostar Combined With Chemotherapy Followed by Endostar Maintenance Therapy to Treat Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: NSCLC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Jinsheng Ren, Simcere Pharmaceutical Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM090801
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — endostar protein; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar with chemotherapy (Experimental): All eligible patients will receive Endostar in combination with Gemcitabine plus Platinum-based chemotherapy for 4 cycles (21 days for each cycle). Endostar treatment will continue after completion of chemotherapy cycles until disease progression.
  Interventions: Drug: Endostar; Drug: Gemcitabine-Cisplatin chemotherapy

INTERVENTIONS:
Drug: Endostar — 7.5mg/m2/day, iv, from day 1 to day 14
  Other Names: Recombinant Human Endostatin Injection
Drug: Gemcitabine-Cisplatin chemotherapy — Gemcitabine 1000 mg/m2, iv, on day 1, 8 Cisplatin 80mg/m2, iv, on day 1, 2, 3
  Other Names: GP chemotherapy

SUMMARY:
This single arm study will assess the safety and efficacy of Endostar combined with chemotherapy (Gemcitabine plus Platinum-based chemotherapy) followed by Endostar maintenance therapy in patients with stage IIIB/IV non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
All eligible patients will receive Endostar in combination with Gemcitabine plus Platinum-based chemotherapy for 4 cycles (21 days for each cycle). Endostar treatment will continue after completion of chemotherapy cycles until disease progression. Efficacy will be evaluated every two cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of inoperable stage IIIB/IV NSCLC
* At least one measurable lesion
* Age of 18-75 years
* Life expectancy > 3 months
* ECOG performance status 0-2
* Adequate hematologic, renal, and hepatic function

Exclusion Criteria:

* Prior systemic chemotherapy for NSCLC
* Evidence of any unstable diseases (serious infection, grade 4 hypertension, unstable angina, congestive heart-failure, compromised renal or hepatic function, nonhealing wound or bone fracture)
* Concurrent anticoagulation therapy
* Evidence of bleeding diathesis or coagulopathy
* Pregnant or lactating women
* Allergic to E.coli preparation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | July 2011

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | July 2011
Clinical Benefit Response (CBR) | July 2011
Overall Survival (OS) | July 2011
Survival Rate | one year
Adverse Events | July 2011

CONTACTS AND LOCATIONS:
Overall Officials: Yiping Zhang, Dr., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China